CLINICAL TRIAL: NCT04698655
Title: Influence of Osteoarthritis eDucational Information and General Practitioner Endorsement on ExerCISe IntentiONs, Beliefs and Willingness to Exercise: the DECISION Randomised Controlled Trial.
Brief Title: Influence of Osteoarthritis Information on Treatment Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Belinda Lawford, Principal Investigator, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20744
Record Dates: First submitted 2020-12-13; First posted 2021-01-07 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Education; Decision aid; Beliefs
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Asked to read a single-A4 page of brief osteoarthritis information ("what is osteoarthritis")
  Interventions: Other: Information on osteoarthritis
- Treatment options group (Experimental): Asked to read brief osteoarthritis information + two A4 pages of information on treatment options ("osteoarthritis treatment options")
  Interventions: Other: Information on treatment options; Other: Information on osteoarthritis
- Treatment options + recommendation group (Experimental): Asked to read brief osteoarthritis information + information on treatment options + receive hypothetical general practitioner recommendation for exercise
  Interventions: Other: Information on treatment options; Other: Recommendation from general practitioner; Other: Information on osteoarthritis

INTERVENTIONS:
Other: Information on treatment options — Asked to read two A4 pages of information on treatment options ("osteoarthritis treatment options")
  Arms: Treatment options + recommendation group; Treatment options group
Other: Recommendation from general practitioner — Receive a hypothetical general practitioner recommendation for exercise
  Arms: Treatment options + recommendation group
Other: Information on osteoarthritis — Asked to read 1 A4 page of brief information on osteoarthritis

SUMMARY:
The aim of this study is to evaluate the effect of educational information, with and without a general practitioner recommendation to exercise, on willingness to undertake exercise/physical activity for knee osteoarthritis. Eligible participants will be aged 45+ years and will not currently have osteoarthritis, knee pain, or any condition that makes them unable to exercise. Participants will be asked to complete an online survey, during which they will be randomised to one of three groups and shown different types of educational information to read. Outcome measures will be collected as part of the survey before and after participants read the educational information presented to them.

DETAILED DESCRIPTION:
3-arm superiority online randomised controlled trial (delivered within one survey). Participants will complete an online survey, during which they will be presented with a hypothetical scenario asking them to imagine that they had recently developed knee pain and have gone to see their general practitioner. Participants will then be randomised to one of 3 different groups (described below). Each group will be shown different types of educational material and asked to read the information carefully. Once they have finished reading the material, they will be asked to complete follow-up outcome measures to determine whether their beliefs about osteoarthritis management strategies have changed.

The 3 trial groups are:

I. Control group: asked to read a single-A4 page of brief osteoarthritis information ("what is osteoarthritis"); II. Treatment options group: asked to read brief osteoarthritis information + two A4 pages of information on treatment options ("osteoarthritis treatment options"), and; III. Treatment options + recommendation group: asked to read brief osteoarthritis information + information on treatment options + receive a hypothetical GP recommendation for exercise

ELIGIBILITY:
Inclusion Criteria:

* Aged 45+ years

Exclusion Criteria:

* Been told by a health professional that they have osteoarthritis in any joint/anywhere in the body
* Have experienced any knee pain in the prior 3 months
* Unable to read English
* Have had a joint replacement in any knee or hip joint
* Have any health condition that makes unable to exercise

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Belief that an exercise or physical activity program is the most appropriate management option for their knee | Immediately after reading educational information in survey
  Measured on an 11-point scale (0 = strongly disagree 10 = strongly agree)

SECONDARY OUTCOMES:
Belief surgery, weight loss, x-rays, injections and medications are the most appropriate management options for their knee | Immediately after reading educational information in survey
  Measured on an 11-point scale (0 = strongly disagree 10 = strongly agree)
Intentions to request a referral to an orthopedic surgeon, physiotherapist, and dietitian or to request prescription for medications, an injection, and an x-ray for their knee | Immediately after reading educational information in survey
  Measured on an 11-point scale (0 = definitely would not 10 = definitely would)
Belief about the effectiveness of surgery, weight loss, x-rays, injections and medications for people with knee osteoarthritis | Immediately after reading educational information in survey
  Measured on an 11-point scale (0 = strongly disagree 10 = strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda J Lawford, Principal Investigator — University of Melbourne
Locations (1):
- The University of Melbourne, Carlton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No